CLINICAL TRIAL: NCT07331857
Title: First-in-Human Pilot Study for the Evaluation of Digma Medical's Endoscopic Gastrointestinal Ablation Device (EGAD) in the Esophagus
Brief Title: Digma System First in Human (FIH) Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Digma Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLD-014-BE
Record Dates: First submitted 2025-12-05; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Barrett's Esophagus (BE)
Keywords: endoscopic gastrointestinal ablation device (EGAD); Barrett's esophagus (BE); esophagus; Digma V2 System; First-in-human pilot study
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Intervention Model Description: Prospective, open-label, single-arm, early feasibility study (EFS) in 2 Patient cohorts.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endoscopic Gastrointestinal Ablation Device (EGAD) (Experimental): Application of different doses of laser energy in the ablation of esophageal mucosa using the Digma System and the EGAD procedure (Cohort A) followed by application of the optimal dose for treatment of patients with BE with LGD or HDG without a visible lesion (Cohort B).
  Interventions: Device: Endoscopic Gastrointestinal Ablation Device (EGAD)

INTERVENTIONS:
Device: Endoscopic Gastrointestinal Ablation Device (EGAD) — Application of different doses of laser energy in the ablation of esophageal mucosa using the Digma System and the EGAD procedure (Cohort A) followed by application of the optimal dose for treatment of patients with BE with LGD or HDG without a visible lesion (Cohort B).

SUMMARY:
Prospective, open-label, single-arm, early feasibility study (EFS) in 2 Patient cohorts: Cohort A - Dose finding / Dose response study in patients with various etiologies undergoing Esophagectomy and Cohort B - Patients with Barrett's Esophagus (BE) with Low-Grade Dysplasia (LDG) or High-Grade Dysplasia (HGD) without a visible (excisable) lesion. This is a pilot study which plan to enroll up to 5 eligible patients in the First Cohort (A) and up to 15 patients in the Second Cohort (B) of the study.

DETAILED DESCRIPTION:
Study intervention means tha application of different doses of laser energy in the ablation of esophageal mucosa using the Digma System and the Endoscopic Gastrointestinal Ablation Device (EGAD) procedure (Cohort A) followed by application of the optimal dose for treatment of patients with BE with Low-Grade Dysplasia (LGD) or High-Grade Dysplasia (HDG) without a visible lesion (Cohort B).

EGAD is a proprietary, controlled laser ablation system for the treatment of endoluminal pathologies of the gastrointestinal tract. EGAD achieves high precision through a unique optical design that controls laser energy, beam size, wavelength, and focal plane. This allows for effective ablation that is limited to the mucosa of pre-selected regions of interest, avoiding a wider and deeper injury to healthy tissue. EGAD procedure can be performed safely in a standard endoscopy suite under direct endoscopic visualization. In this First-in-Human pilot feasibility study, we plan to assess the feasibility of EGAD for achieving mucosal ablation (1) in healthy esophageal tissue in patients undergoing esophagectomy for esophageal cancer or other indications (Barrett's mucosa may be ablated as well) - Cohort A; and (2) In patients with Barrett's Esophagus with low and/or high-grade dysplasia (BORN = Barrett´s Oesophagus-Related Neoplasia) without a visible (excisable) lesion - Cohort B.

ELIGIBILITY:
Inclusion Criteria:

Cohort A:

1. Male or Female ≥18 years of age at the time of consent.
2. Scheduled to undergo esophagectomy for malignant or benign indications .
3. Contain enough healthy (or with BE) tissue to be ablated (≥1cm) by for EGAD treatment.
4. Capable of providing written informed consent.

Cohort B:

1. Male or Female ≥18 and ≤ 70 years of age at the time of consent.
2. Documented diagnosis of Barrett's Esophagus (BE) with LGD or HGD, confirmed by biopsy specimen analysis.
3. No visible lesion in the esophagus (suitable for endoscopic resection).
4. Scheduled to undergo Endoscopic eradication therapy (EET) procedure of Barrett's Esophagus (BE) with dysplasia.
5. BE affected tissue length ≥1 cm and ≤ 5cm (as measured endoscopically).
6. Capable of providing written informed consent.
7. Willingness and ability to comply with follow-up requirements, including endoscopies and biopsies.
8. Ability to tolerate and take oral proton pump inhibitor (PPI) medication.

Exclusion Criteria:

Cohort A:

1. Severe medical comorbidities that preclude esophagectomy.
2. Any medical or technical condition that may preclude endoscopy during surgical esophagectomy at the discretion of operating surgeon.
3. Any previous procedures involving esophageal tissue resection or ablation.
4. Patients with incomplete healing of tissue following radiation at the area-of-interest.
5. Subjects undergoing (or having undergone) photodynamic therapy.
6. Subjects of high surgical risk, in which any delay in the esophagectomy surgery may, in the option of the PI, increase the risk for to Adverse event (AE) / Serious Adverse event (SAE).
7. Presence of esophageal stricture preventing passage of the endoscope or investigational catheter .
8. Any anatomical abnormality (such as but not limited to, esophageal dilation) that, at the discretion of the investigator may preclude the laser ablation.
9. Presence of esophageal varices in the esophagus.
10. Presence of severe bleeding or severe inflammation at the time of endoscopy of EGAD.
11. Female who is pregnant, breast-feeding or intends to become pregnant or is of childbearing potential and not using an adequate contraceptive method .
12. Any disorder, which in the investigator's opinion might jeopardize participant's safety or compliance with the Clinical Investigation Plan (CIP).
13. Patient refusal or inability to provide written informed consent.

Cohort B:

1. Severe medical comorbidities that preclude endoscopy or multiple co-morbidities placing the patient at risk or otherwise unsuitable for trial participation .
2. Previous radiotherapy in the chest.
3. Previous Endoscopic Mucosal resection (EMR) / Endoscopic Submucosal Dissection (ESD) in the esophagus.
4. Subjects currently undergoing or subject that had previous ablative therapy within the esophagus (e.g., Photodynamic Therapy (PDT), Multipolar Electrocoagulation (MPEC), Argon Plasma Coagulation (APC), laser treatment, radiofrequency ablation (RFA).
5. Presence of esophageal stricture preventing passage of the endoscope or investigational catheter .
6. Active esophagitis.
7. Esophageal or gastric varices.
8. Subject diagnosed with portal hypertension.
9. Subject diagnosed with Liver cirrhosis.
10. Presence of severe bleeding or severe inflammation in the area-of-interest.
11. Use of anticoagulants or antiplatelet agents that cannot be discontinued 5 days prior to the procedure
12. Active systemic infection or malignancy.
13. History of esophagectomy
14. History of locally advanced (>T1a) esophageal cancer treated endoscopically/by chemoradiotherapy.
15. Subjects with known coagulation conditions (e.g. uncontrolled coagulopathy)
16. Concurrent chemotherapy.
17. Female who is pregnant, breast-feeding or intends to become pregnant or is of childbearing potential and not using an adequate contraceptive method.
18. Any disorder, which in the investigator's opinion might jeopardize participant's safety or compliance with the CIP .
19. Patient refusal or inability to provide written informed consent.
20. Known history of unresolved drug or alcohol dependency that would limit ability to comprehend or follow instructions, uncontrolled psychiatric illness (including recent inpatient psychiatric treatment, psychosis, moderate to severe depression, illicit substance abuse) or any psychiatric diagnosis which in the opinion of the investor would preclude participation in the study.
21. Concurrent enrollment in an investigational drug or device trial that clinically interferes with study endpoints.
22. Subject that is unwilling or unable to comply with study visits and other study procedures as required per protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Cohort A: Incidence of severe immediate adverse events (AEs) | Day 1, ESOPHAGECTOMY surgery
  Cohort A: Incidence of severe immediate adverse events (AEs) that are directly associated with EGAD procedure (esophageal perforation, bleeding, patient hemodynamic or respiratory decompensation during the procedure or death following the procedure).
Cohort B: Incidence of immediate severe AE | Day 1
  Cohort B: Incidence of immediate severe AE (including esophageal perforation, bleeding, patient hemodynamic or respiratory decompensation during the procedure or death following the procedure, esophageal stricture rate after ablation).
Cohort B: Incidence of late severe AE | 10-12 months follow-up, following each visit and procedure
  Cohort B: Incidence of late severe AE (including esophageal perforation, bleeding, patient hemodynamic or respiratory decompensation during the procedure or death following the procedure, esophageal stricture rate after ablation). A dedicated designed Questioner will be used.
Cohort A: Dose response effects of ablation on mucosal tissue | Day 1, ESOPHAGECTOMY surgery
  Cohort A: Dose response effects of ablation on mucosal tissue (assessed by histopathological assessment of mucosal eradication (coagulation necrosis).
Cohort B: Eradication of dysplasia level and of visible segment of BE | 10-12 months follow-up, at each follow-up visit
  Cohort B: Eradication of dysplasia level and of visible segment of BE assessed macroscopically.

SECONDARY OUTCOMES:
Adverse events related to the procedure (Cohort A+B) | Day 1
  Incidence of any adverse events related to the procedure.
Maximal ablation depth (cohort A) | Day 1, ESOPHAGECTOMY surgery
  Evaluation of maximum ablation depth. Grading of histology to be conducted in accordance with accepted histological score grading such as depicted in van Munster SM et al. Endoscopy 2021,53,1162-1168 wherein thermal injury was semi-quantitatively scored and the proportion of tissue injury was calculated (depth of thermal changes / total tissue thickness).
Maximal ablation volume (cohort A) | Day 1, ESOPHAGECTOMY surgery
  Evaluation of maximum ablation volume. Following esophagectomy, all resected ablated tissue will be submitted for histopathologic analysis. Analysis of the EGAD treatment ablation sites for evaluation of the ablation outcomes (such as extent of mucosal ablation and depth of penetration) will be conducted per a predefined histological protocol and criterium.
Dose response effect of treatment(s) on depth-of-penetration. (cohort A) | Day 1, ESOPHAGECTOMY surgery
  Evaluation of the dose-dependent effect of treatment on penetration depth, examining how different intensities or doses of the therapy used affect the extent to which the treatment penetrates the tissue, in order to assess the relationship between dose, efficacy, and the potential risks of excessive treatment. Grading of histology to be conducted in accordance with accepted histological score grading such as depicted in van Munster SM et al. Endoscopy 2021,53,1162-1168 wherein thermal injury was semi-quantitatively scored and the proportion of tissue injury was calculated (depth of thermal changes / total tissue thickness).
Assessment of collateral impact as assessed by histopathologic evaluation. | 10-12 months follow-up or when eradication of BE is achieved
  Assessment of secondary effects, in which histopathological examination is used to assess the extent of undesirable changes in tissues outside the target area in order to determine whether the procedure has caused damage to surrounding structures or other unforeseen tissue reactions.
Rate of complete eradication of dysplasia (cohort B) | 10-12 months follow-up
  The degree of complete eradication of dysplasia, which assesses the extent to which all dysplastic changes in the mucosa have been completely removed or replaced by normal epithelium after treatment, in order to evaluate the overall effectiveness of the therapy and minimize the risk of persistent or recurrent precancerous lesions.
Rate of eradication of intestinal metaplasia. (cohort B) | 10-12 months follow-up
  The degree of eradication of intestinal metaplasia, which monitors how much of the pathologically altered mucosa has been successfully removed or replaced by normal epithelium after treatment in order to assess the effectiveness of therapy and the likelihood of long-term remission.
Eradication of macroscopically visible segment of BE. | 10-12 months follow-up
  Eradication of macroscopically visible Barrett's esophagus, in which complete removal of all clearly altered mucosal areas is assessed to ensure that the pathological epithelium has been treated in its entirety and that no residual focal changes remain.
Assessments of lesion ablation - safe margin area. | 10-12 months follow-up
  Evaluation of lesion ablation, focusing primarily on the size and consistency of the safety margin to ensure that the treated area sufficiently exceeds the boundaries of the lesion and minimizes the risk of incomplete removal.
Assessment of technical aspects of the procedure-time | Day 1
  Evaluation of the technical time of the procedure (minutes or hours), assessing in particular the time required.

CONTACTS AND LOCATIONS:
Overall Officials: Shlomit Chappel-Ram, BSc,PhD, Study Director — Digma Medical General Manager
Locations (1):
- Fakultní nemocnice u sv. Anny v Brně, Gastroenterologické a hepatologické oddělení, Brno, Czechia

IPD SHARING:
Plan to Share IPD: No
All information concerning this study that was not previously published is considered confidential information. This confidential information shall remain the sole property of Digma Medical Ltd.; it shall not be disclosed to others without written consent of Digma Medical Ltd. and shall not be used except in the performance of this study (see also Clinical Trial Agreement). Any investigator involved with this study is obligated to provide the Sponsor with complete test results and all data derived from the study.